CLINICAL TRIAL: NCT03595072
Title: Assessment of Effect of Vagal Nerve Stimulator (VNS) on Electrocorticograms Recorded by Responsive Neurostimulator (RNS) in Patients With Drug Resistant Epilepsy
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty securing funding due to COVID-19
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-0578
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stimulation: patient ECOG recordings during active VNS stimulation
  Interventions: Other: observation of VNS stimulation effects
- interstimulation: the same patient ECOG during inter-stimulation periods

INTERVENTIONS:
Other: observation of VNS stimulation effects — ECOGs will be recorded during VNS stimulation and inter stimulation periods
  Groups: Stimulation

SUMMARY:
This study will investigate whether a Vagal Nerve Stimulator (VNS) causes measurable desynchronization and reduces epileptiform activity, such as spikes and seizures, in electrocorticograms (ECOGs) recorded by a Responsive Neurostimulator (RNS) in patients who have both devices implanted.

Specific aims of the study:

1. Evaluate the change in frequency of epileptiform discharges during active VNS stimulation compared to interstimulation baseline periods
2. Evaluate the change in frequency of seizures during active VNS stimulation compared to interstimulation baseline periods
3. Evaluate the change in the number of RNS activations during active VNS stimulation compared to interstimulation baseline periods
4. Evaluate the change in synchronization of background ECoG (electrocorticogram) during VNS stimulation compared to interstimulation baseline periods.

DETAILED DESCRIPTION:
Drug resistant epilepsy, is defined by the International League Against Epilepsy (ILAE) as "the failure of adequate trials of two tolerated and appropriately chosen and used AED (Antiepileptic drug) schedules (whether as monotherapies or in combination) to achieve sustained seizure freedom." About a third of epilepsy cases are drug resistant and are considered for non-pharmacologic treatment. Surgical removal (resection) of the seizure focus is the treatment of choice in drug resistant epilepsy with focal onset. However, curative surgery is not always feasible, e.g. if it would lead to unacceptable deficits, or if there are seizure onset areas in both sides of the brain. In addition, depending on the circumstances, patients treated with surgery do not become seizure free in about 10-80% of cases, depending on presence or absence of a lesion and location of the seizure focus. Other surgical options include implantation of neuromodulatory devices, such as Vagus Nerve Stimulator (VNS) and Responsive Neurostimulator (RNS).

IIa. Vagus Nerve Stimulator (VNS) Brain surgery was the only surgical option for some patients in this drug-resistant patient population until 1997 when the VNS was approved by the FDA. VNS is approved for use as an adjunctive therapy in reducing the frequency of seizures in adults and adolescents over age 12 diagnosed with medically refractory partial onset seizures (FDA 1997). The vagus nerve and its centers (nuclei) in the brainstem have, in general, an inhibitory effect on organs. VNS therapy can suppress seizures by sending mild pulses of electrical energy to the vagus nerve in regular intervals. The default setting of stimulation are cycles of 30-seconds "on" and 5-minutes "off". These stimulation pulses are supplied by a thin, round battery-containing device which is placed under the skin on the left side of the chest, like a pacemaker, with wires connecting the generator to the vagus nerve on the left side of the neck. VNS is not likely to stop seizures (seizure freedom rate with VNS added range from 2-9%), but it provides a ~50% chance of cutting the seizure frequency in half (Ben-Menachem 1999, Scherrmann 2001,Morris 1999, Kuba 2009).

IIb. Responsive Neurostimulator (RNS) The RNS was FDA approved in 2013. The RNS System provides responsive cortical stimulation through an implanted programmable neurostimulator connected to depth and/or subdural cortical strip leads targeted to the seizure focus. The RNS device continually monitors brain activity (electrocorticography [ECoG]). It is programmed by the physician to detect seizure patterns and provide appropriate electrical stimulation within a few seconds of the seizure onset. RNS was approved by the FDA for use as an adjunctive therapy in reducing the frequency of seizures in individuals 18 years of age or older with partial (focal) onset seizures who have undergone diagnostic testing that localized to no more than two epileptogenic foci, are refractory to two or more antiepileptic medications, and currently have frequent and disabling seizures (FDA 2013). The generator of the device is implanted in the patient's skull and wires connect to the leads in or on the brain (see Figure 2). Depending on where in the brain it is implanted, RNS is associated with seizure free intervals of 6 months in 26-29% of patients and of 12 months in 14-15% of cases. The rate of seizure freedom is relatively low, compared to resections, but the chance of a marked (~70%) seizure reduction is high (Geller 2017, Jobst 2017).

IIc. No studies to date have investigated the effect of VNS stimulation on the more recently FDA approved RNS. The initial RNS feasibility study listed VNS as an exclusion criteria as it was not clear how the two devices would interact. However, before RNS was available, patients with a seizure focus or several foci that could not be surgically removed, were implanted with VNS. Therefore, in the current post-approval phase of RNS treatment, many patients already have a VNS which has not brought the hoped for seizure relief. Across centers it has been standard practice to implant RNS in patients who have a VNS, and to keep the VNS turned on, if the patient reported clinical benefit. Even though there are no guidelines, the rationale for not removing a VNS before RNS implantation appears to be as follows:

1. The devices are not linked or physically close together and are not enabled to communicate with each other.
2. Current delivered by either device penetrates only targeted tissue in the immediate vicinity of the electrodes and is not able to reach the other device.
3. Each device provides a different mechanism of action and is a separate, independent modality to influence seizures, similar to medications and VNS being different therapy modalities that act in a complementary fashion.
4. To date, no case of a concerning interaction has been described.

Thus, many patients with drug-resistant epilepsy have both VNS and RNS implanted. So far, the investigators have no data and no knowledge of how the VNS influences brain activity, as recorded by RNS, close to a seizure focus. The presence of continually-recording Intracranial RNS electrodes provides a unique opportunity to study changes in normal and abnormal ECoG patterns during VNS stimulation.

III. PRELIMINARY STUDIES/PROGRESS REPORT:

VNS continues to be used as an adjunctive therapy as many patients with drug resistant epilepsy are either opposed to a resection or the invasive surgery required for RNS implantation, or are not a good candidate for these surgeries based on location and/or number of epileptogenic foci. VNS was approved by the FDA in 1997 for use as an adjunctive therapy in reducing the frequency of seizures in adults and adolescents over age 12 diagnosed with medically refractory partial onset seizures. Data suggests that only 2-9% (Ben-Menachem 1999, Scherrmann 2001) of patients become seizure free after implantation, but over time 43-49% of patients experience a >50% drop in seizure frequency (Morris 1999; Kuba 2009.)

In the RNS comparative study - which investigated device efficacy - seizure frequency was measured for 3 months in both the Treatment Group (received stimulation) and the Control Group (did not receive stimulation). The Treatment Group had a reduction in seizures of 37.9% and the Control Group had a reduction in seizures of 17.3%. Seizure frequency was also measured by determining the number of patients who achieved a 50% reduction in seizures. After 1 year, almost half of the patients in the treatment group (44%) had at least 50% fewer seizures. And at 2 years, over half of the patients (55%) had at least 50% fewer seizures. Seven-year follow-up showed up to 70% seizure reduction, and up to 15% of patients reported seizure free periods of 12 months (Geller et al 2017, Jobst et al 2017).

VNS was an exclusion criterion in the RNS clinical trial to avoid any interference of the devices. Of all patients enrolled in the study, 32% had previously used VNS without sufficient benefit (Bergey 2015). This patient population had the VNS explanted in order to participate in the RNS trial. Nowadays, after approval of the device, 27% of patients who receive a RNS also have a VNS (unpublished data collected by Neuropace® the company manufacturing the device, personal communication). In clinical practice, there is no contraindication to combined neurostimulation using VNS in addition to RNS.

To date, no head-to-head comparison studies have been done that compare efficacy of RNS compared to VNS.

The effect of VNS stimulation on the RNS recordings (ECoGs) will be determined during one clinic visit scheduled for RNS assessment and interrogation. ECoGs with brain activity during VNS stimulation and in-between stimulation - baseline - intervals will be recorded, stored, and later analyzed. During this visit, as an exception to standard of care, the regular, patient-specific VNS "on-" and "off-times" will be turned off and VNS stimulation will be triggered by the investigator using a magnet that activates the VNS for the set time of 30 seconds (see detailed protocol below.) This will represent a temporary change in a patient's VNS settings for the time of the recordings, but at the end of the visit, the stimulation "on" and "off" times, will be returned to the previous home settings. These VNS changes are unlikely to affect the patient's seizure control, as VNS effect on seizures is a result of months and years of stimulation. Though, just like at home, the patient is expected to feel the VNS "on-time" as a sensation in the throat, often described as "tickling", which may prompt clearing the voice or a cough, as well as a transient hoarseness.

A stimulation time of 30 seconds was chosen for stimulation duration as the typical default setting for VNS stimulation is 30 seconds and many patients are treated at default settings. A period of 30 seconds before and after stimulation was chosen as recording time to allow for at least 1 min between stimulations which is standard of care. Since the purpose of this study is to compare the effect of active VNS stimulation on the brain and ECoG to intervals without VNS stimulation, the investigators chose timing that would allow for maximum number of stimulations/recordings within a clinic appointment that is within the standard of care in terms of frequency of stimulations

D. DETAILED PROTOCOL FOR RESEARCH DATA COLLECTION IN CLINIC:

1. RNS recording equipment (so-called "wand") used to connect to the device through the skin and collect data will be secured to the patient's scalp over the implanted RNS computer. This will be done using a velcro cap provided by the RNS Manufacturer (NeuroPace®). Connection will be made with device and real-time ECoG data visualized on laptop. Clinic appointment will proceed as per standard of care.

1a. Electromyography (EMG) electrode will be in place over left side of neck close to the VNS contacts. This electrode will be able to detect muscle signal and artifact related to VNS stimulation which will confirm successful VNS activation when triggered.

2. VNS will be interrogated using a handheld interrogation device. Stimulation parameters will be recorded and output current will be turned to zero. VNS magnet stimulation duration will be set to 30 seconds (rationale, see above) with pulse width and output current at the patient's baseline stimulation settings. All settings will be within accepted ranges for standard of care.

3. ECoG recording will be initiated on laptop, by turning on "Real-time ECoG"

4. Thirty seconds into the recording, the VNS will be triggered with magnet stimulation which will produce a 30-second vagus nerve stimulation ("stim"). 30 seconds later, the recording will be stopped and stored.

4a. This will generate a 30 sec pre-stim, a 30 sec stim, and a 30 sec post-stim recording.

5. This will be repeated 30 times per patient for a total of 30 VNS stimulations or up to 45 minutes of patient time

6. At the end of the appointment, VNS will be returned to its scheduled stimulations with any adjustments needed as would be part of standard of care.

ELIGIBILITY:
INCLUSION CRITERIA:

1. A patient of the University of Colorado Hospital Epilepsy clinic;
2. Have had either VNS and/or RNS implanted;
3. Age 18 years to 75 years.

EXCLUSION CRITERIA:

1. Not capable of making a medical decision;
2. Unable to comprehend study details, or
3. Unable to adequately communicate secondary to intellectual or language barrier.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a pilot study which plans to enroll all current patients with both VNS and RNS with potential to enroll further participants as more patients have both devices implanted.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of epileptiform discharges during active VNS stimulation and during interstimulation baseline periods | 1 day of clinic appointment
Change in frequency of seizures during active VNS stimulation and during interstimulation baseline periods | 1 day of clinic appointment
Change in the number of RNS activations during active VNS stimulation and during interstimulation baseline periods | 1 day of clinic appointment
Change in synchronization of background ECoG (electrocorticogram) during VNS stimulation. | 1 day of clinic appointment

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Destefano, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver | Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No